CLINICAL TRIAL: NCT04458597
Title: Stereotactic Pelvic Adjuvant Radiation Therapy in Cancers of the Uterus: A Phase 1 Pilot Study (SPARTACUS)
Brief Title: Stereotactic Pelvic Adjuvant Radiation Therapy in Cancers of the Uterus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPARTACUS
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Endometrioid Adenocarcinoma; Serous Carcinoma; Clear Cell Carcinoma; Carcinosarcoma; Dedifferentiated Carcinoma
MeSH Terms: conditions — Carcinoma, Endometrioid; Cystadenocarcinoma, Serous; Adenocarcinoma, Clear Cell; Carcinosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Image-guided adjuvant pelvic radiotherapy — Image-guided adjuvant pelvic radiotherapy delivered at an SBRT prescription dose of 30 Gy in 5 fractions if feasible, well-tolerated and effective for the adjuvant treatment of high-risk endometrial cancer.

SUMMARY:
Advanced technology has enabled radiation oncologists to more accurately and precisely target radiation to areas at risk while maximally sparing healthy tissue. Furthermore, there is growing evidence demonstrating both safety and efficacy for SBRT. We propose that these advantages are translatable to the adjuvant treatment of endometrial cancer. We submit that a prescription dose of 30 Gy in 5 fractions, which equates to a 2 Gy equivalent dose (i.e an EQD2) (α/β = 10 Gy) of 48 Gy, compares favorably to the EQD2 delivered standardly for adjuvant treatment (44.25 Gy via 45Gy/25Fx; 50 Gy at vaginal surface for vault brachytherapy) and therefore should be effective and safe dose in the adjuvant setting. Through precision delivery and careful dosimetry the treatment should be safe and well tolerated with minimal impact on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who have undergone hysterectomy for curative intent, with histologically confirmed endometrioid adenocarcinoma, serous or clear cell carcinoma, or carcinosarcoma or dedifferentiated carcinoma
* Patient is a candidate for adjuvant pelvic radiation (+/- vault brachytherapy), meeting one of the following conditions:

  * High grade histology OR
  * Outer-half myometrial invasion and FIGO grade 1-2 OR
  * FIGO stage II - IIIC1 (all gross nodal disease must be resected)
* Patient is willing and able to give informed consent to participate in this clinical trial.
* Age ≥18 years.
* Patients who are to receive adjuvant systemic therapy in addition to pelvic radiotherapy will be eligible provided that there is at minimum a 3-week interval between any radiation treatment and chemotherapy treatments. Adjuvant systemic therapy may be given before or after radiation treatment.
* Patient must be willing and able to complete the QLQ-C30 questionnaire with EN-24 companion as described in the study protocol.
* Primary language of the patient must be English or, if a patient's primary language is not English, they are still able to participate provided the QLQ-C30 and EN-24 is available in their primary language.

Exclusion Criteria:

* Patient has had prior pelvic radiotherapy.
* Patient has received neo-adjuvant systemic therapy
* Patient has a contraindication to pelvic radiotherapy, such as but not limited to a connective tissue disease or inflammatory bowel disease.
* Patient has a contraindication to iodinated CT contrast.
* Patient has a hip prosthesis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Assess the acute urinary and bowel toxicities | Baseline to 2 years post-treatment.
  Acute urinary and bowel toxicities associated with adjuvant SBRT treatment in the setting of high-risk endometrial cancer will be assessed using the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: David D'Souza, M.D., Principal Investigator — London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada